CLINICAL TRIAL: NCT03560908
Title: Dasatinib Combined With Multi-agents Chemotherapy in Relapsed t(8;21) Acute Myeloid Leukemia With KIT D816 Mutation
Brief Title: Dasatinib Combined With Chemotherapy in Relapsed t(8;21) Acute Myeloid Leukemia With KIT D816 Mutation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No enough eligable participants enrolled
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2018004
Record Dates: First submitted 2018-06-01; First posted 2018-06-18 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2020-03

CONDITIONS: Relapsed AML; T(8;21); C-KIT Mutation
Keywords: leukemia,myeloid, acute; relapse; mutation; KIT; dasatinib
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dasatinib plus chemotherapy (Experimental): Dasatinib combined with chemotherapy for relapsed t(8;21) AML with D816 mutation
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Dasatinib 70mg twice a day will be administered orally for 2 weeks along with re-induction chemotherapy from day 1 of chemotherapy. Recommended re-induction regimens include (1)FLAG: Fludarabine 30mg/m2/d,d1-5;cytarabine 1g-2g/m2/d,d1-5;±G-CSF;(2)IA/DA:idarubicin 8-12mg/m2/d,d1-3 or daunorubicin 45-60mg/m2/d，d1-3;cytarabine 100-200mg/m2/d，d1-7;(3)CAG:Aclarubicin 20mg/d,d1-4；cytarabine 15mg/m2/Q12h,d1-14; ±G-CSF.The chemotherapy regimen is not limited to recommended regimens. Patients will be recommended to receive allogeneic hematopoietic stem cell transplantation (HSCT) once complete remission is achieved. Otherwise, they will continue the consolidation chemotherapy.

SUMMARY:
In this multi-center, open-label, no control,prospective clinical trial, a total of 30 relapsed acute myeloid leukemia with t(8;21) translocation and KIT D816 mutation patients will be enrolled. Dasatinib 70 mg twice a day will be administrated for two weeks from day 1 of re-induction chemotherapy. The purpose of current study is to determine the clinical efficacy and tolerability of combination therapy of dasatinib with multi-agent chemotherapy in relapsed acute myeloid leukemia with t(8;21) translocation and KIT D816 mutation.

ELIGIBILITY:
Inclusion Criteria:

1. T(8;21)acute myeloid leukemia patients with KIT D816 mutation diagnosed by bone marrow morphology, immunology, molecular genetics. The diagnosis and classification are according to WHO 2016 criteria.
2. Conform to relapsed diagnosis.Only morphological relapsed cases will be enrolled.Molecular relapsed and isolated extramedullary relapsed cases are not eligible.
3. Age is not limited. Both male and female are eligible.
4. Eastern Cooperative Oncology Group performance status (ECOG-PS):0-2 point.
5. Informed consent form must be signed by patients themselves before enrolled for patients aged 18 years or older. Informed consent form must be signed by the legal guardian for patients younger than 18 years.

Exclusion Criteria:

1. Patients with other blood diseases at the same time (such as haemophilia, primary myelofibrosis and so on) are not considered suitable.
2. Isolated extramedullary relapsed leukemia.
3. With other malignant tumors accompanied with AML and needed treatment. 4 .Patients who are unsuitable for the trial considered by investigators.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
composite complete remission (CR) rate | 8 weeks
  confirmed rate of complete remission (CR) plus complete remission with incomplete blood count(CRi)

SECONDARY OUTCOMES:
mortality during induction chemotherapy | 30 days
  all deaths from start of chemotherapy
post relapsed overall survival | 2 years
  2 years overall survival from the date of relapse
overall survival | 5 years
  5 years overall survival from the date of diagnosis
post relapsed disease free survival | 2 years
  2 years disease free survival from the date of new complete remission

CONTACTS AND LOCATIONS:
Overall Officials: Jianxiang Wang, Dr., Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- HBDH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided